CLINICAL TRIAL: NCT05681741
Title: Impact of Cardiopulmonary Bypass Flow on Cerebral Autoregulation in Cardiac Surgery, a Cross-over Study
Brief Title: Impact of Cardiopulmonary Bypass Flow on Cerebral Autoregulation
Acronym: FLOWMAPCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Sauvegarde (Other)
Collaborators: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Principal Investigator, Johanne Beuvelot, Principal Investigator, Clinique de la Sauvegarde
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Ramsay Sante Sauvegarde Clinic
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Autoregulation; Cardiopulmonary Bypass; Mean Arterial Pressure
Keywords: FlowMapca

STUDY DESIGN:
Intervention Model Description: parallel affectation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- current pump flow (between 2 and 2.4 l/min/m²) (Sham Comparator): the pump flow will be constant during this randomized phase
  Interventions: Procedure: current versus high pump flow
- high pump flow (between 2.6 and 3 l/min/m²) (Active Comparator): the pump flow will be constant during this randomized phase
  Interventions: Procedure: current versus high pump flow

INTERVENTIONS:
Procedure: current versus high pump flow — during each phase of randomized pump flow, arterial pressure will be increased from 40 to 90 mmHg with vasodilators and/or vasoconstrictors

SUMMARY:
Cerebral autoregulation is defined by the capacity of the brain to maintain a constant cerebral blood flow (CBF) despite variations of arterial pressure. However, when the arterial pressure is below a critical threshold, cerebral blood decreases.

This critical threshold is called the lower limit of cerebral autoregulation (LLA).

Cardiopulmonary bypass is a unique environment wherein systemic blood flow is totally controlled by the cardiopulmonary bypass pump. High pump flows combined with low arterial pressures has been shown to not compromise neurologic postoperative outcomes.

Our hypothesis is that that LLA may depend on the cardiopulmonary bypass flow, ie the LLA may decrease when the cardiopulmonary bypass flow increases, explaining why low arterial pressure may be well tolerated.

DETAILED DESCRIPTION:
Cerebral tissue perfusion is partly ensured by cardiac output and arterial pressure. In cardiac surgery, and especially during bypass surgery, one of the main objectives is to maintain sufficient blood flow and an optimal mean arterial pressure (MAP) to limit the deleterious consequences of organ hypoperfusion. To have a physiological regional organ blood flow, some organs, such as the brain, need a minimum MAP threshold (the lower limit of autoregulation, LLA) to ensure a constant cerebral blood flow (CBF). This is known as the cerebral autoregulation (CA). As the brain is at high risk of ischemia and definitive functional consequences in case of cerebral hypoperfusion, maintaining MAP above the LLA of the brain limit the deleterious postoperative neurological outcome.

CA can be determined by continuously calculating the correlation between MAP and CBF. CBF is assessed by continuous monitoring of the middle cerebral artery velocity (mV). moving Pearson correlation coefficient between 30 consecutive, paired MAP and cerebral blood flow velocity values will be calculated to generate the mean velocity index (Mx). The Blood pressure in the autoregulation range is indicated by an Mx value that approaches zero (there is no correlation between flow velocity and MAP), whereas an Mx approaching 1 indicates dysregulated cerebral blood flow (flow velocity and MAP are correlated). A value of 0.4 is accepted as the threshold of CA corresponding to the LLA.

During cardiopulmonary bypass (CPB), MAP is physiologically related to bypass flow and systemic vascular resistance. The adjustment of MAP during CPB is therefore achieved by the administration of vasoconstrictors or vasodilators as well as by the variations of the pump flow.

This research assumes that a change in the pump flow rate will lead to a change in the LLA. Therefore, if the flow rate is higher, it is possible that the LLA will be lower.

In this randomized trial, two different rates of pump flow will be compared with respect to LLA testing.

Regional brain oxygen saturation, assessed by near-infrared spectroscopy will also be monitored during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over the age of 18
* Patient scheduled to undergo valvular heart surgery with planned CPB
* Patient with a Euroscore below 7%
* Patient affiliated or entitled to a social security scheme
* Patient having received informed information about the study and having signed a free and informed consent to participate in the study

Exclusion Criteria:

* Patient with untreated or uncontrolled severe hypertension despite treatment
* Patient with chronic renal failure, with glomerular filtration < 30 mL/min/1.73m² or requiring a kidney transplant
* Patient with left ventricular ejection fraction < 40%
* Patient with a history of ischemic stroke
* Patient having or about to benefit from renal vascular surgery
* Patient with preoperative sepsis
* Patient who required a norepinephrine infusion within 24 hours before surgery
* Patient presenting with an inaccessible temporal Doppler window
* Patient candidate for emergency surgery
* Pregnant, parturient or breastfeeding woman
* Patient with preoperative uni or bilateral carotid stenosis > 50%
* Protected patient: adult under guardianship, curators or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
measurement of MAP LLA (mmHg) | 15 to 25 min during the procedure
  Determination of MAP LLA according to the calculation of the mean velocity index

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Desebbe, MD, Principal Investigator — Clinique de la Sauvegarde
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No